CLINICAL TRIAL: NCT00825539
Title: A Single-dose, Placebo-controlled, Stratified, Randomized, Double-blind, Crossover to Study Pharmacodynamic Effects of AQW051 Followed by a 4-week Multiple-dose Safety and Tolerability in People With Chronic Stable Schizophrenia.
Brief Title: Pharmacodynamic/Pharmacokinetic Study of AQW051 in Schizophrenia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CAQW051A2202
Record Dates: First submitted 2009-01-19; First posted 2009-01-21 (Estimated); Last update posted 2020-12-24 (Actual); Status verified 2013-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Manic depression; anxiety
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Anxiety Disorders | interventions — 3-(6-p-tolylpyridin-3-yloxy)-1-azabicyclo(2.2.2)octane

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- AQW051 (Experimental)
  Interventions: Drug: AQW051

INTERVENTIONS:
Drug: AQW051
  Arms: AQW051
Drug: Placebo
  Arms: Placebo

SUMMARY:
Part 1 of the study will assess the enhancement of task-related brain activation (BOLD response) in key brain areas in schizophrenia during the performance of working memory, episodic memory and visual activation tasks as measured by functional magnetic resonance imaging (fMRI) in people with schizophrenia. Part 2 of the study will assess the safety and tolerability of multiple doses of AQW051 in people with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of schizophrenia according to the Diagnostic and Statistical Manual of Mental Disorders IV (DSM IV/DSM IV TR)
2. Subjects will be currently treated with the stable regimen of one or more of the following second generation antipsychotics: olanzapine, risperidone, paliperidone, quetiapine, ziprasidone, aripiprazole.
3. Subjects will meet the following symptom criteria:

   * Brief Psychiatric Rating Scale (BPRS) Hallucinatory Behavior or Unusual Thought Content item scores less than or equal to 5
   * BPRS Conceptual Disorganization item score less than or equal to 4
   * Simpson-Angus Scale (SAS) total score less than or equal to 6
   * Calgary Depression Scale (CDS) total score less than or equal to 10
4. Subjects will meet the following cognitive performance criteria:

   * Maximum performance level: Performance below 1.0 SD from perfect performance on the Hopkins Verbal Learning Test (HVLT) total (31 or less),
   * Minimum performance level: subject must be able to validly complete the fMRI cognitive paradigms
   * WTAR: 5th grade reading level assessment
5. Subjects must be symptomatically stable and not suffer from an acute exacerbation of their psychosis
6. Female subjects of childbearing potential must be using two acceptable methods of contraception, (e.g., intra-uterine device plus condom, spermicidal gel plus condom, diaphragm plus condom, etc.), from the time of screening and for the duration of the study, through study completion. Pregnancy tests are required of all female subjects regardless of reported sterilization.

   When performed at screening and practice visit, the result of this test must be received before the subject may be dosed.
7. Male subjects must be using two acceptable methods of contraception, (e.g., spermicidal gel plus condom) for the entire duration of the studyuntil the Study Completion visit.
8. Subject must have sufficiently stable overall health, as determined by the Investigator. The regular intake of concomitant drugs will be allowed, if the patient is on stable treatment for at least 3 months prior to study enrollment and the concomitant drug does not belong to the list of medication that are not allowed according to Appendix 3. If the patient takes more than one concomitant medication, it is at the Investigator's discretion to decide about the patient's eligibility, depending on the nature of the concomitant medications and the patient's overall health.

Exclusion criteria:

1. Current treatment with conventional antipsychotics (e.g. fluphenazine, haloperidol) or clozapine
2. Current treatment with an anticholinergic or other agent known to adversely interfere with the cholinergic system
3. Subjects with a DSM-IV diagnosis of substance abuse (other than nicotine) within the last month.
4. Subjects with a history of significant head injury/trauma, as defined by:

   * Loss of consciousness (LOC) for more than 1 hour
   * Recurring seizures resulting from the head injury
   * Clear cognitive sequelae of the injury
   * Cognitive rehabilitation following the injury
5. Subjects with a medical or neurological disorder or treatment for such disorder that could interfere with the study medication of the assessment of the subject
6. Use of certain concomitant medication

No grapefruit or grapefruit juice is to be consumed for 14 days prior to dosing until 7 days following the last dose.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2009-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Part 1: Assess BOLD response in key brain areas in schizophrenia patients during the performance of tasks as measured by (fMRI) in people with schizophrenia. | 2 years (Part 1: 1 year)
Part 2: Assess safety and tolerability of multiple doses of AQW051 schizophrenia patients. | Part 2: 8 months

SECONDARY OUTCOMES:
Measure: To assess the effects of a single dose of AQW051 on performance of working and episodic memory tasks in people with schizophrenia. (Part 1) | Time Frame: 2 years (Part 1: 1 year; Part 2: 8 months)
Measure: To determine the relationship of exposure to brain activation after a single dose of AQW051 in people with schizophrenia. (Part 1) | 2 years (Part 1: 1 year; Part 2: 8 months)
Measure: To determine the dose-exposure response relationship of multiple doses of AQW051 in people with schizophrenia. (Part 2) | 2 years (Part 1: 1 year; Part 2: 8 months)
Measure: To explore effects of multiple doses of AQW051 on measures of cognition in people with schizophrenia. (Part 2) | 2 years (Part 1: 1 year; Part 2: 8 months)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- United States (7):
  - West LA VA Healthcare Center (UCLA), Los Angeles, California
  - Department of Psychiatry & Behavioural Sciences, Feinberg School of Medicine (Northwestern University), Chicago, Illinois
  - Maryland Psychiatric Research Centre, Spring Grove Hospital Grounds, Baltimore, Maryland
  - Massachusetts General Hospital (Freedom Trail Clinic), Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Columbia University, New York, New York
  - JUH Clinical Research (Duke University),, Butner, North Carolina

REFERENCES:
- [Derived] Barch DM, Marder SR, Harms MP, Jarskog LF, Buchanan RW, Cronenwett W, Chen LS, Weiss M, Maguire RP, Pezous N, Feuerbach D, Lopez-Lopez C, Johns DR, Behrje RB, Gomez-Mancilla B. Task-related fMRI responses to a nicotinic acetylcholine receptor partial agonist in schizophrenia: A randomized trial. Prog Neuropsychopharmacol Biol Psychiatry. 2016 Nov 3;71:66-75. doi: 10.1016/j.pnpbp.2016.06.013. Epub 2016 Jun 28. PMID 27371157
- See also: Results for CAQW051A2202 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=10383